CLINICAL TRIAL: NCT02570750
Title: Non-interventional Study Of The Effect Of Smoking Status Of The Patient On The Success Of Etanercept Therapy In Psoriasis
Brief Title: The Effect Of Smoking Status Of The Patient On The Success Of Etanercept Therapy In Psoriasis
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801392
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Results first posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-06

CONDITIONS: Chronic Plaque Psoriasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: smokers patients group: smokers (more than 10 cigarettes per day)
  Interventions: Behavioral: QUESTIONNAIRE ON SMOKING HABITS
- Group 2 : non-smokers patients group: Smoking status will be classified as current and never/former. Former smokers will be defined as those who had stopped smoking at least 1 year before being interviewed for this study
  Interventions: Behavioral: QUESTIONNAIRE ON SMOKING HABITS

INTERVENTIONS:
Behavioral: QUESTIONNAIRE ON SMOKING HABITS — Data on smoking will include the age at which cigarette smoking began and ceased and the average amount smoked daily. Intensity (number of cigarettes smoked per day), duration of smoking (years), and time since cessation (years) will be categorized. Also, the smoking status of the patient prior psoriasis diagnosis will be assessed (smoker or non-smoker and years of smoking prior to psoriasis diagnosis).
  Smoking habit evaluation: baseline and changes in smoking habit at 12 and 24-weeks follow-up time points.

SUMMARY:
The main purpose of this study is to assess the effect of smoking status on the success of Etanercept therapy in patients with moderate-to-severe psoriasis.

DETAILED DESCRIPTION:
Study hypothesis was based on the following rationale:

* Psoriasis vulgaris is a chronic inflammatory skin disease with several extracutaneous manifestations and significant comorbidities (among others cardiovascular disease, metabolic syndrome, obesity and depression).
* An increased prevalence of smoking among psoriasis patients, as compared with healthy subjects, has been observed in several studies
* More recent studies suggest that cigarette smoking may trigger the development of psoriasis through oxidative, inflammatory and genetic mechanisms.Furthermore, smoking is associated with the clinical severity of psoriasis
* Smoking also contributes to higher morbidity and mortality from smoking related disorders in these patients There is now some evidence that patients with psoriasis who smoke tend to be less responsive to treatment

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years at the time of screening
* Clinical diagnosis of chronic plaque type psoriasis for at least 6 months as determined by the subjects medical history, and confirmation of the diagnosis through physical examination by the investigator
* Patients who are scheduled by their dermatologist to initiate treatment with Etanercept prescribed independently by the investigator as per local clinical practice guideline
* Stable plaque psoriasis for at least 2 months prior to Baseline
* Diagnosis of severe psoriasis defined as PASI > 10
* Eligible for Etanercept treatment according to Summary of Product Characteristics (SmPC)
* Smokers with smoking >10 cigarettes daily for smokers group (Group 1) or non-smokers for non-smoking group (Group 2)
* Evidence of a personally signed and dated informed consent form indicating that the subject has been informed of all pertinent aspects of the study

Exclusion Criteria:

* Previous or current treatment with antipsoriatic biologic drugs, such as Etanercept, infliximab, adalimumab, ustekinumab, alefacept, efalizumab.
* Exclusion Criteria according to the Enbrel® SmPC, with particular attention to: hypersensitivity to the active substance (etanercept) or to any of the excipients; sepsis or risk of sepsis, active infections, including chronic or localised infections.
* Positive pregnancy test, breast feeding or considering becoming pregnant during the study
* Clinically significant drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with severe plaque psoriasis and starting an anti-TNF treatment with etanercept
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2016-12-05 (Actual); Study Completion 2016-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- Romania (29):
  - Bratianu Diagnostic and Treatment Center Pitesti / Dermatology Department, Piteşti, Argeş
  - County Emergency Hospital Pitesti / Dermatology Department, Piteşti, Argeş
  - SCBI Ambulatory Cluj-Napoca / Dermatology Department, Cluj-Napoca, Cluj
  - Dr. Remus Orasan Medical Office, Cluj-Napoca, Cluj
  - Dr Ianosi Medical Center Craiova / Dermatology Department, Craiova, Dolj
  - Emergency County Hospital Craiova / Dermatology Department, Craiova, Dolj
  - Helios Medica Ambulatory Craiova / Dermatology Department, Craiova, Dolj
  - County Hospital Targoviste / Dermatology Department, Târgovişte, Dâmbovița County
  - Hospital for Infectious Diseases Dermatovenereology and Psychiatry Baia Mare / Dermatology Departmen, Baia Mare, Maramureş
  - County Emergency Hospital Drobeta Turnu Severin / Dermatology Department, Drobeta-Turnu Severin, Mehedinți County
  - Derma Luxury Style Medical Office - DR. Serban Diana Ramona Reghin, Reghin, Mureș County
  - Sighisoara Municipal Hospital / Dermatology Department, Sighișoara, Mureș County
  - Mures County Clinical Hospital / Dermatology Department, Târgu Mureş, Mureș County
  - County Emergency Hospital Ploiesti / Dermatology Department, Ploieşti, Prahova
  - County Emergency Hospital Zalau / Dermatology Department, Zalău, Sălaj County
  - Municipal Emergency Hospital Timisoara / Dermatology Department, Timișoara, Timiș County
  - County Emergency Hospital "Saint Pantelimon" Focsani / Dermatology Department, Focşani, Vrancea
  - Stoica Dan Marius Dermatology Office Arad, Arad
  - Emergency Hospital Bacau / Dermatology Department, Bacau
  - County Emergency Hospital "Mavromati" Botosani / Dermatology Department, Botoșani
  - County Emergency Hospital Brasov / Dermatology Department, Brasov
  - Emergency Hospital Militar Central "Dr. Carol Davila" Bucharest / Dermatology Department, Bucharest
  - Elias Emergency University Hospital Bucharest / Dermatology Department, Bucharest
  - Ambulatory Railway Hospital No. 2 Bucharest / Dermatology Department, Bucharest
  - Clinical Hospital Colentina Bucharest / Dermatology Department, Bucharest
  - Hospital "Dr. Victor Babes" Bucharest / Dermatology Department, Bucharest
  - County Emergency Hospital "Saint Spiridon" Iasi / Dermatology Department, Iași
  - Railways Hospital Iasi / Dermatology Department, Iași
  - Bucovina Medical Office Suceava, Suceava

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801392&StudyName=Non-interventional%20Study%20Of%20The%20Effect%20Of%20Smoking%20Status%20Of%20The%20Patient%20On%20The%20Success%20Of%20Etanercept%20Therapy%20In%20Psoriasis

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Non Smokers: Non-smoker participants (defined as those who never smoked or quitted smoking at least 1 year prior to the enrollment in study) diagnosed with moderate to severe plaque psoriasis and who were eligible for initiating the etanercept treatment based on physician's discretion as per summary of product characteristics (SmPC), were observed prospectively in this study for 24 weeks. According to SmPC, recommended dose for etanercept is 25 milligram (mg) twice weekly, 50 mg once weekly or 50 mg twice weekly as subcutaneous injection.
- Etanercept: Smokers: Smoker participants (defined as those who smoke more than 10 cigarettes per day), diagnosed with moderate to severe plaque psoriasis, and who were eligible for initiating the etanercept treatment based on physician's discretion as per SmPC, were observed prospectively in this study for 24 weeks. According to SmPC, recommended dose for etanercept is 25 mg twice weekly, 50 mg once weekly or 50 mg twice weekly as subcutaneous injection.
Period: Overall Study
Arm/Group | Etanercept: Non Smokers | Etanercept: Smokers
Started | 110 | 73
Completed | 96 | 68
Not Completed | 14 | 5
Not completed — Inclusion/exclusion criteria deviation | 1 | 0
Not completed — Protocol deviation | 4 | 2
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Population: Per protocol set included all treated participants.
Groups:
- Etanercept: Non Smokers: Non-smoker participants (defined as those who never smoked or quitted smoking at least 1 year prior to the enrollment in study) diagnosed with moderate to severe plaque psoriasis and who were eligible for initiating the etanercept treatment based on physician's discretion as per SmPC, were observed prospectively in this study for 24 weeks. According to SmPC, recommended dose for etanercept is 25 mg twice weekly, 50 mg once weekly or 50 mg twice weekly as subcutaneous injection.
- Total: Total of all reporting groups
Arm/Group | Etanercept: Non Smokers | Etanercept: Smokers | Total
Number analyzed (Participants) | 96 | 68 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (13.5) | 49.1 (14.5) | 51.0 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 31 | 69
  Male | 58 | 37 | 95

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Psoriasis Assessment and Severity Index (PASI) Score at Week 24
Description: PASI is the combined assessment of lesion severity and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Body divided into 4 sections (head and neck [h], arms [u], trunk [t], legs [l]); each area scored by itself and scores combined for final PASI score. For each section, percent body surface area (A) of skin involved was estimated on a scale of 0 (no involvement) to 6 (90-100 percent involvement), severity was estimated by clinical signs: erythema (E), induration (I), scaling (S) on a 5 point scale: 0 (no involvement) to 4 (very marked involvement). Final PASI = sum of severity parameters for each section*area score*weighing factor (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4).
Time Frame: Baseline, Week 24
Population: Per protocol set included all treated participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: Non Smokers | Etanercept: Smokers
Number analyzed (Participants) | 96 | 68
units on a scale
  Baseline | 23.1 (6.2) | 23.4 (6.1)
  Change at Week 24 | 16.5 (5.2) | 17.1 (5.4)

2. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI)
Description: The DLQI was a 10-item questionnaire that measures the impact of skin disease on participant's quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. The DLQI total score ranges from 0 (not at all) to 30 (very much): 0-1 = no effect at all on the participant's life; 2-6 = small effect on the participant's life; 7-12 = moderate effect on the participant's life; 13-18 = very large effect on the participant's life; 19-30 = extremely large effect on the participant's life. Higher scores indicate more impact on quality of life of participants.
Time Frame: Baseline, Week 12, 24
Population: Per protocol set included all treated participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: Non Smokers | Etanercept: Smokers
Number analyzed (Participants) | 96 | 68
units on a scale
  Baseline | 22.0 (5.3) | 21.7 (4.8)
  Change at Week 12 | 12.3 (6.0) | 12.8 (4.9)
  Change at Week 24 | 16.4 (6.0) | 16.8 (4.6)

3. Secondary Outcome: Percentage of Participants With Psoriasis Area and Severity Index 75 (PASI75) Response at Week 12 and 24
Description: PASI is the combined assessment of lesion severity and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Body divided into 4 sections (head and neck [h], arms [u], trunk [t], legs [l]); each area scored by itself and scores combined for final PASI score. For each section, percent body surface area (A) of skin involved was estimated on a scale of 0 (no involvement) to 6 (90-100 percent involvement), severity was estimated by clinical signs: erythema (E), induration (I), scaling (S) on a 5 point scale: 0 (no involvement) to 4 (very marked involvement). Final PASI = sum of severity parameters for each section*area score*weighing factor (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4). PASI75 response was defined as at least a 75 percent (%) reduction in PASI relative to baseline.
Time Frame: Week 12, 24
Population: Per protocol set included all treated participants.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept: Non Smokers | Etanercept: Smokers
Number analyzed (Participants) | 96 | 68
percentage of participants
  Week 12 | 9.3 | 4.4
  Week 24 | 45.8 | 44.1

4. Secondary Outcome: Percentage of Participants With Psoriasis Area and Severity Index 50 (PASI50) Response at Week 12 and 24
Description: PASI is the combined assessment of lesion severity and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Body divided into 4 sections (head and neck [h], arms [u], trunk [t], legs [l]); each area scored by itself and scores combined for final PASI score. For each section, percent body surface area (A) of skin involved was estimated on a scale of 0 (no involvement) to 6 (90-100 percent involvement), severity was estimated by clinical signs: erythema (E), induration (I), scaling (S) on a 5 point scale: 0 (no involvement) to 4 (very marked involvement). Final PASI = sum of severity parameters for each section*area score*weighing factor (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4). PASI50 response was defined as at least a 50% reduction in PASI relative to baseline.
Time Frame: Week 12, 24
Population: Per protocol set included all treated participants.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept: Non Smokers | Etanercept: Smokers
Number analyzed (Participants) | 96 | 68
percentage of participants
  Week 12 | 77.0 | 82.3
  Week 24 | 97.9 | 98.5

5. Secondary Outcome: Change From Baseline in Psoriasis Assessment and Severity Index (PASI) Score at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: Per protocol set included all treated participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: Non Smokers | Etanercept: Smokers
Number analyzed (Participants) | 96 | 68
units on a scale | 12.6 (4.4) | 12.8 (4.6)

6. Secondary Outcome: Change From Baseline in Psoriasis Assessment and Severity Index (PASI) Score in Obese Participants
Description: PASI is the combined assessment of lesion severity and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Body divided into 4 sections (head and neck [h], arms [u], trunk [t], legs [l]); each area scored by itself and scores combined for final PASI score. For each section, percent body surface area (A) of skin involved was estimated on a scale of 0 (no involvement) to 6 (90-100 percent involvement), severity was estimated by clinical signs: erythema (E), induration (I), scaling (S) on a 5 point scale: 0 (no involvement) to 4 (very marked involvement). Final PASI = sum of severity parameters for each section*area score*weighing factor (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4). Participants who had bone marrow index >30 kilogram per meter square were said to be obese in this outcome measure.
Time Frame: Baseline, Week 12, 24
Population: Per protocol set included all treated participants. Here, "N" (overall number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: Non Smokers | Etanercept: Smokers
Number analyzed (Participants) | 36 | 10
units on a scale
  Baseline | 24.2 (6.12) | 23.9 (7.14)
  Change at Week 12 | 12.2 (4.52) | 12.1 (5.21)
  Change at Week 24 | 17.1 (5.79) | 16.8 (4.26)

ADVERSE EVENTS:
Time Frame: Baseline up to 1 year
Description: Same event may appear as both an adverse event and serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Adverse events data was planned to be reported for overall population.
Arm/Group | Etanercept: Non Smokers | Etanercept: Smokers
All-Cause Mortality (participants affected / at risk) | 0/96 | 1/68
Serious Adverse Events (participants affected / at risk) | 2/96 | 3/68
Other Adverse Events (participants affected / at risk) | 4/96 | 4/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept: Non Smokers (N=96) | Etanercept: Smokers (N=68)
Inflammation at site injection (Infections and infestations) | 0 | 1
Diabetic gangrene (Endocrine disorders) | 1 | 0
Cerebellar haematoma (Nervous system disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erytrodermic psoriasis (Immune system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept: Non Smokers (N=96) | Etanercept: Smokers (N=68)
Erytrodermic psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Injection site erythema (General disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Increase of serum transaminases (Investigations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.